CLINICAL TRIAL: NCT00279799
Title: HIV Prevention Maintenance for African American Teens
Brief Title: HIV Prevention for African American Teens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ralph J. DiClemente, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00041131; NIMH 5 R01 MH070537-08
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-09

CONDITIONS: Sexually Transmitted Diseases
Keywords: Sexually Transmitted Diseases, HIV, condom use, adolescents
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Afiya group intervention + HIV prevention phone sessions (Experimental): Afiya group-based intervention plus individually tailored HIV prevention phone sessions
  Interventions: Behavioral: Afiya HIV Prevention Intervention
- Afiya group session + nutrition phone sessions (Active Comparator): Afiya group-based intervention plus individually tailored nutrition phone sessions
  Interventions: Behavioral: Afiya HIV prevention intervention

INTERVENTIONS:
Behavioral: Afiya HIV Prevention Intervention — Group-based session plus individually tailored HIV prevention phone sessions
  Arms: Afiya group intervention + HIV prevention phone sessions
Behavioral: Afiya HIV prevention intervention — Afiya group-based intervention + nutrition phone sessions (attention control)
  Arms: Afiya group session + nutrition phone sessions

SUMMARY:
AFIYA aims to reduce both the risk of Sexually Transmitted Infections (STIs) and HIV in young African American females through a culturally and gender appropriate intervention (group sessions) coupled with an individualized HIV Telephone Maintenance Intervention.

DETAILED DESCRIPTION:
African-American adolescent females are a population at high risk for HIV infection. Recent findings suggest that culturally and gender appropriate HIV educational programs can significantly reduce sexual risk behaviors among this vulnerable population over the short term. It is unclear as to whether these programs have long-term effects. Thus, the aim of this project is to develop and test a culturally and gender-appropriate sexual health education program designed to promote long-term maintenance of HIV preventive sexual behaviors over a long follow-up period.

700 African-American female adolescents' between the ages of 14-20 will be enrolled in this trial. Adolescents will be recruited from youth currently seeking services at several family planning clinics in Atlanta, Georgia. Adolescents who are eligible and willing to participate in the project will complete an initial ACASI survey. The survey is designed to assess adolescents' sexual risk and preventive behaviors. Biological specimens are collected and tested for common STI's. Free DOT (Directly Observed Therapy) is provided through the clinics. Urine pregnancy screens will also be conducted. After they complete the assessment, adolescents will receive a sexual health education program that was developed by the Principal Investigator. This program (HORIZONS) has been shown to be effective in reducing sexual risk behaviors over the short-term. Trained African American female health educators will deliver the sexual health education program. Adolescents will then be assigned, by chance alone, to one of two groups: one group will get periodic telephone contacts designed to reinforce sexual health promotion and the other group will get periodic telephone contacts that promote healthy dietary practices. Thus, while all adolescents receive the same sexual health education program, half will get telephone calls emphasizing sexual health and half will get an equal number of telephone calls emphasizing nutritional health.

The primary aims of the proposed project are:

Primary Aim 1. To determine whether adding a telephone educational component to a sexual health education program will reduce incident STD infection over a 36-month follow-up.

Primary Aim 2. To determine if adding a telephone educational component to a sexual health education program can maintain HIV-preventive behaviors.

We will ask adolescents to come back to participating clinics to complete follow-up assessments at 6 months, 12-months,18-months, 24-months, 30-months and 36-months after completing the initial assessment. We will test the effects of adding the telephone sexual health educational program to maintain or enhance adolescents' use of HIV prevention behaviors and reduce incident STDs. If successful, the findings could have important implications for HIV prevention.

ELIGIBILITY:
Inclusion Criteria:

* Female; African American; age 14-20; receiving care at participating clinic;report having unprotected vaginal sex in last 6 months; ability to give written informed consent

Exclusion Criteria:

* pregnant or trying to get pregnant; married; any condition that would preclude attending group-based intervention sessions.

Ages: 14 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 701 (Actual)
Dates: Start 2005-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Incident STD infection, particularly chlamydial infections, confirmed by laboratory PRC testing over a 36 month follow-up. | 36 months post-randomization.

SECONDARY OUTCOMES:
Proportion of condom-protected vaginal sex acts and sex while high or drunk over the 36 month follow-up. | 36 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J DiClemente, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Fulton County Department of Health and Wellness, Atlanta, Georgia
  - Grady Hospital Teen Clinic, Atlanta, Georgia
  - Planned Parenthood of GA, Atlanta, Georgia

REFERENCES:
- [Background] DePadilla L, Windle M, Wingood G, Cooper H, DiClemente R. Condom use among young women: modeling the theory of gender and power. Health Psychol. 2011 May;30(3):310-9. doi: 10.1037/a0022871. PMID 21553975
- [Background] Sales JM, Latham TP, Diclemente RJ, Rose E. Differences between dual-method and non-dual-method protection use in a sample of young African American women residing in the Southeastern United States. Arch Pediatr Adolesc Med. 2010 Dec;164(12):1125-31. doi: 10.1001/archpediatrics.2010.230. PMID 21135341
- [Background] Sales JM, Lang DL, DiClemente RJ, Latham TP, Wingood GM, Hardin JW, Rose ES. The mediating role of partner communication frequency on condom use among African American adolescent females participating in an HIV prevention intervention. Health Psychol. 2012 Jan;31(1):63-9. doi: 10.1037/a0025073. Epub 2011 Aug 15. PMID 21843001
- [Background] Sales JM, Brown JL, Diclemente RJ, Davis TL, Kottke MJ, Rose ES. Age differences in STDs, sexual behaviors, and correlates of risky sex among sexually experienced adolescent African-American females. J Pediatr Psychol. 2012 Jan-Feb;37(1):33-42. doi: 10.1093/jpepsy/jsr076. Epub 2011 Sep 20. PMID 21933811
- [Background] Diclemente RJ, Young AM, Painter JL, Wingood GM, Rose E, Sales JM. Prevalence and correlates of recent vaginal douching among African American adolescent females. J Pediatr Adolesc Gynecol. 2012 Feb;25(1):48-53. doi: 10.1016/j.jpag.2011.07.017. Epub 2011 Nov 3. PMID 22051790
- [Background] Brown JL, Sales JM, Diclemente RJ, Latham Davis TP, Rose ES. Characteristics of African American adolescent females who perceive their current boyfriends have concurrent sexual partners. J Adolesc Health. 2012 Apr;50(4):377-82. doi: 10.1016/j.jadohealth.2011.07.008. Epub 2011 Sep 23. PMID 22443842
- [Background] Sales JM, DiClemente RJ, Brody GH, Philibert RA, Rose E. Interaction between 5-HTTLPR polymorphism and abuse history on adolescent African-American females' condom use behavior following participation in an HIV prevention intervention. Prev Sci. 2014 Jun;15(3):257-67. doi: 10.1007/s11121-013-0378-6. PMID 23479192
- [Derived] DiClemente RJ, Wingood GM, Sales JM, Brown JL, Rose ES, Davis TL, Lang DL, Caliendo A, Hardin JW. Efficacy of a telephone-delivered sexually transmitted infection/human immunodeficiency virus prevention maintenance intervention for adolescents: a randomized clinical trial. JAMA Pediatr. 2014 Oct;168(10):938-46. doi: 10.1001/jamapediatrics.2014.1436. PMID 25155070
- [Derived] Swartzendruber A, Sales JM, Brown JL, Davis TL, DiClemente RJ, Rose E. Predictors of repeat Chlamydia trachomatis and/or Neisseria gonorrhoeae infections among African-American adolescent women. Sex Transm Infect. 2013 Feb;89(1):76-82. doi: 10.1136/sextrans-2012-050530. Epub 2012 Dec 12. PMID 23236082